CLINICAL TRIAL: NCT01972022
Title: A Prospective Optical Coherence Tomography (OCT) Study on Coronary Vessel Wall Response to Stent Eluting Everolimus From a Biodegradable Polymer (EES SYNERGY™) Compared With Stent Eluting Zotarolimus From a Durable Polymer (ZES, RESOLUTE Integrity™).
Brief Title: TRANSFORM OCT TRiple Assessment of Neointima Stent FOrmation to Reabsorbable polyMer With Optical Coherence Tomography
Acronym: TRANSFORM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Responsible Party: Principal Investigator, GGuagliumi, MD, A.O. Ospedale Papa Giovanni XXIII
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRANSFORM 1207/2013
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-03

CONDITIONS: Coronary Artery Lesions
Keywords: Drug Eluting Stents; Bioabsorbale Polymer Coating; Neoatherosclerosis; Stent Coverage; Stent Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EES SYNERGY™ (Experimental): coronary artery lesions treated with Bioabsorbable Polymer EES
  Interventions: Device: EES SYNERGY™
- ZES, RESOLUTE Integrity™ (Active Comparator): coronary artery lesions treated with ZES, RESOLUTE Integrity™ stent system
  Interventions: Device: ZES, RESOLUTE Integrity™

INTERVENTIONS:
Device: EES SYNERGY™ — percutaneous coronary intervention with implantation of Bioabsorbable Polymer EES
  Arms: EES SYNERGY™
Device: ZES, RESOLUTE Integrity™ — percutaneous coronary intervention using ZES, RESOLUTE Integrity™ coronary stent
  Arms: ZES, RESOLUTE Integrity™

SUMMARY:
First prospective randomized controlled study to evaluate in an 'all-comers' population with coronary artery disease whether treatment with a novel everolimus eluting stent (EES) with a biodegradable polymer is superior to a durable polymer zotarolimus eluting stent (ZES), with respect to the long term vascular response to treatment These data are important to ascertain the superiority of a new generation DES with bioabsorbable polymer coating to reduce the long term development of in-stent neoatherosclerosis.

DETAILED DESCRIPTION:
During the last decade a considerable clinical experience has been accumulated with the use of drug eluting coronary stents with durable polymers, that permanently cover the metallic stent scaffold, allowing the local delivery of anti-restenotic agents. However durable polymers have been associated with an increased risk of late and very late stent thrombosis and the anticipated development of in stent neo-atherosclerosis. Since permanent polymer coatings may have pro-inflammatory effects, with delayed healing and prolonged endothelial dysfunction, current research on DES has focused on the use of biodegradable polymer coatings, which disappear after a short period of drug-release (3-4 months). Current clinical guidelines recommend at least 6-12 months of dual antiplatelet therapy (DAPT) after DES implantation,in order to prevent ST. Recent data obtained by pooled analyses of ZES, support a significant reduction of the DAPT to the same range used with bare metal stents. The substantial delays in DES healing observed from multiple human pathology series and in-vivo studies using Optical Coherence Tomography (OCT) were not assessed as risk factors for prolonged used of DAPT. However different patient cohorts might have different responses to stent implantation. In addition, there is no comparative evidence on long term development of neo-atherosclerosis in bioabsorbable versus permanent polymer DES. OCT allows precise assessment of stent strut apposition and coverage and accurate measures of different tissue components of neoatherosclerosis. This study is the first attempting to characterize the early and late vascular responses to novel bioabsorbable polymer EES (SYNERGY™) compared with a permanent polymer benchmark novel generation ZES (RESOLUTE INTEGRITY™) .The stent comparator has been selected due to the large use across the interventional cardiology community and the recent approval from European Regulators Authorities to update the CE (Conformité Européenne) mark labeling to only one-month duration of dual anti-platelet therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years of age;
2. Subject has stable angina or acute coronary syndrome (including acute myocardial infarction) with evidence of coronary ischemia and de novo atherosclerotic coronary artery disease in multiple vessels with an indication for stent implantation;
3. Target lesion stenosis is ≥ 70% (visual estimate)
4. All target lesions require treatment with stents having diameters from 2.25 mm to 4.0 mm (visual estimate)
5. Target lesion length ≥10 mm and ≤50 mm for each target lesion(s)
6. Subject must sign Ethics Committee approved informed consent prior to undergoing any study specific procedure;
7. Subject must be willing and able to comply with specified follow-up schedule.

Exclusion Criteria:

1. Unprotected left main coronary disease;
2. Chronic total occlusion;
3. Severe calcified target lesion(s) which cannot be, in the investigator's opinion, successfully treated;
4. Significant angulation in the target vessel that, in the Investigator's opinion, may preclude stent delivery and deployment;
5. Bifurcation disease involving a side branch ≥ 2.5 mm in diameter;
6. Restenotic lesions;
7. Target lesion(s) within a coronary bypass graft (e.g., saphenous vein or arterial graft);
8. In the Investigator's opinion, the lesion is not suitable for stenting or OCT imaging (e.g. extreme tortuosity, very distal lesions).
9. Documented left ventricular ejection fraction ≤30%;
10. Serum creatinine > 2.0 mg/dl at the time of treatment;
11. Recipient of heart transplant;
12. Subject with malignancies or other comorbidities (i.e. severe liver, renal, pulmonary, pancreatic disease) with life expectancy less than 18 months or that may results in protocol non-compliance;
13. Known bleeding or hyper-coagulable disorder;
14. Known allergy to stent components or any antiplatelet recommended drug
15. Planned medical or surgical procedures requiring modification of DAPT regimen within 3 months after the index procedure;
16. Women of childbearing potential without negative pregnancy test within 7 days before enrollment
17. Currently participating in an investigational study that has not completed the primary endpoint or that clinically interferes with the study endpoints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-03 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
percentage of frames with in stent-lipid laden neointima, neovascularization, calcification and thin-cap fibro-atheroma (TFCA) | 18 months
  OCT finding of neoatherosclerosis, counted as percentage of frames with in stent-lipid laden neointima, neovascularization, calcification and thin-cap fibro-atheroma (TFCA) (18 month primary end-point)
length of consecutive frames with uncovered struts | 3 and 18 months
  OCT derived maximum length of consecutive frames with uncovered struts in the two stent arms at 3 and 18 month (3 month primary end-point and 18 months co-primary end-points)

SECONDARY OUTCOMES:
percent well apposed struts at implant without neointima | 3 and 18 months
  OCT derived proportion of well apposed struts at implant without neointima (% uncovered struts) at 3 and 18 months
Acquired stent malapposition | 3 and 18 moths
  Number and extent (max area-volume) of newly acquired malapposed struts at 3 and 18 months.
OCT derived abnormal intraluminal tissue | 3 and 18 months
  Presence of any abnormal intraluminal protruding mass at 3 and 18 months
percentage OCT frames with uncovered struts | 3 and 18 months
  Number/percentage of OCT frames with > 30% uncovered struts at 3 and 18 months
Neointimal tissue thickness | 3 and 18 months
  OCT calculated thickness of tissue covering stents at 3 and 18 months
OCT derived percentage of frames with mature neointima | 3 and 18 months
  Percentage of frames with evidence of mature neointimal coverage in the two stent arms
OCT derived tissue heterogeneity in neointima deposition | 3 and 18 moths
  Segmental tissue heterogeneity in neointima deposition across the entire stent length (as assessed by OCT tissue properties parameters - including normalized intensity, attenuation, tissue contrast) at 3 and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Guagliumi, MD, Principal Investigator — A.O. Papa Giovanni XXIII, Cardiovascular Department
Locations (1):
- A.O. Ospedale Papa Giovanni XXIII, Bergamo, Bergamo, Italy